CLINICAL TRIAL: NCT04488354
Title: A Study to Evaluate the Long-Term Safety of CLBR001, A Lentiviral Based Chimeric Antigen Receptor, In Patients With B-Cell Malignancies Previously Administered CLBR001
Brief Title: Long-term Follow-up Study for Patients Treated With CLBR001 CAR-T
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Calibr, a division of Scripps Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CBR-sCAR19-3002
Record Dates: First submitted 2020-07-20; First posted 2020-07-28 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Relapsed/Refractory B-cell Lymphomas; Diffuse Large B-Cell Lymphoma (DLBCL); Follicular Lymphoma (FL); Chronic Lymphocytic Leukemia (CLL); Marginal Zone Lymphoma (MZL); Mantle Cell Lymphoma (MCL); Small Lymphocytic Lymphoma (SLL); Primary Mediastinal Large B Cell Lymphoma; Transformed Follicular Lymphoma; Waldenstrom Macroglobulinemia; Lymphoplasmacytic Lymphoma; Burkitt Lymphoma
Keywords: CAR-T Cell Therapy; Switchable CAR-T Cell; Autologous Cell Therapy; CD19 Positive Disease; Blood Cancer; Hematological malignancy; Neoplasms; CD19 CAR-T Cell; Long Term Follow Up (LTFU)
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Mantle-Cell; Waldenstrom Macroglobulinemia; Burkitt Lymphoma; Hematologic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CLBR001 treated patients (Experimental): Patients who have been administered with CLBR001
  Interventions: Combination Product: CLBR001 and SWI019

INTERVENTIONS:
Combination Product: CLBR001 and SWI019 — No study drug is administered in this study. Patients who have received CLBR001 autologous CAR-T cells will be evaluated in this trial for long-term safety and efficacy

SUMMARY:
This study is designed as a long-term follow-up study of participants who have receive genetically modified autologous CLBR001 CAR-T cells

DETAILED DESCRIPTION:
Patients will be enrolled following either the completion or early termination/discontinuation from Study NCT04450069 or any protocol in which patients were administered CLBR001. Patients will begin the long-term follow-up period regardless of whether they responded to treatment or progressed on treatment. Patients will be followed for up to 15 years post CLBR001 infusion and will continue to be monitored for safety, immunogenicity, and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* All patients who received at least one CLBR001 cell dose and have either discontinued early or completed the core treatment protocol or any protocol such as a managed access protocol as applicable.
* Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol

Exclusion Criteria:

* There are no specific exclusion criteria for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-01-21 (Actual); Primary Completion 2036-08 (Estimated); Study Completion 2036-08 (Estimated)

PRIMARY OUTCOMES:
Incidence and duration of new adverse events, late onset adverse events, and events of special interest | 15 years
  To measure the incidence and duration of new adverse events, late onset adverse events, and events of special interest
Incidence and duration of new serious adverse events | 15 years
  To measure the incidence and duration of new serious adverse events
Incidence of patients with resolution of adverse events, serious adverse events, and duration that began in previous treatment protocols of CLBR001 | 15 years
  The measure the incidence of patients with resolution of adverse events, serious adverse events, and duration that began in previous treatment protocols of CLBR001
Incidence of new malignancies | 15 years
  The measure the incidence of new malignancies

SECONDARY OUTCOMES:
Overall response | 15 years
  To evaluate clinical efficacy by measuring the overall response by Response Evaluation Criteria In Lymphoma (RECIL) 2017
Duration of response | 15 years
  To evaluate clinical efficacy by measuring the duration of response
Progression free survival | 15 years
  To evaluate clinical efficacy by measuring progression free survival
Proportion of patients undergoing stem cell transplant | 15 years
  To evaluate the proportion of patients undergoing stem cell transplant
Number of CLBR001 CAR+ cells in blood, bone marrow and/or tissue specimens | 3, 6, 9,12 and 24 months
  To measure the number of CLBR001 CAR+ cells in blood, bone marrow and/or tissue specimens
Detectable replication competent lentivirus (RCL) | 15 years
  To measure detectable replication competent lentivirus (RCL)
Titer of anti-drug antibody (ADA) for CLBR001 and SWI019 | 3, 6, 12 months
  To evaluate immunogenicity by measuring the titer of ADA for CLBR001 and SWI019
Duration of detection of ADA for CLBR001 and SWI019 | 3, 6, 12 months
  To evaluate immunogenicity by measuring the duration of detection of ADA for CLBR001 and SWI019

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - City of Hope National Medical Center, Duarte, California
  - University of California at San Diego, San Diego, California
  - University of Chicago, Chicago, Illinois
  - Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Sarah Cannon Research Institute - Tennessee Oncology, Nashville, Tennessee
  - Sarah Cannon Research Institute - Texas Transplant Institute, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rodgers DT, Mazagova M, Hampton EN, Cao Y, Ramadoss NS, Hardy IR, Schulman A, Du J, Wang F, Singer O, Ma J, Nunez V, Shen J, Woods AK, Wright TM, Schultz PG, Kim CH, Young TS. Switch-mediated activation and retargeting of CAR-T cells for B-cell malignancies. Proc Natl Acad Sci U S A. 2016 Jan 26;113(4):E459-68. doi: 10.1073/pnas.1524155113. Epub 2016 Jan 12. PMID 26759369
- [Background] Viaud S, Ma JSY, Hardy IR, Hampton EN, Benish B, Sherwood L, Nunez V, Ackerman CJ, Khialeeva E, Weglarz M, Lee SC, Woods AK, Young TS. Switchable control over in vivo CAR T expansion, B cell depletion, and induction of memory. Proc Natl Acad Sci U S A. 2018 Nov 13;115(46):E10898-E10906. doi: 10.1073/pnas.1810060115. Epub 2018 Oct 29. PMID 30373813